CLINICAL TRIAL: NCT04018248
Title: A Phase I, Open-label, Multi-center, Dose Escalation, and Expansion Study of BR101801 in Adult Patients With Advanced Hematologic Malignancies
Brief Title: BR101801 in Adult Patients With Advanced Hematologic Malignancies(Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BR-101801-CT-101
Record Dates: First submitted 2019-06-14; First posted 2019-07-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Leukemia; B Cell Lymphoma; Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (BR101801): Phase Ia (dose escalation) (Experimental): Patients will receive BR101801 capsules orally, QD in 28-day cycles. The regimen may be changed to BID dosing based on emerging data.
  Interventions: Drug: BR101801 (Phase Ia)
- Treatment (BR101801):Phase Ib (dose expansion) (Experimental): • Subjects with PTCL NOS, PTCL AITL, Nodal PTCL with TFH and PTCL FTCL
  Interventions: Drug: BR101801 (Phase Ib)

INTERVENTIONS:
Drug: BR101801 (Phase Ia) — Phase Ia (dose escalation):25 mg capsules and 100 mg capsules Planned doses are 50, 100, 200, 325, and 450 mg.
  Arms: Treatment (BR101801): Phase Ia (dose escalation)
Drug: BR101801 (Phase Ib) — Phase Ib (dose expansion):25 and 100 mg capsules Doses administered will be determined from Phase Ia data.
  Arms: Treatment (BR101801):Phase Ib (dose expansion)

SUMMARY:
This is a Phase I, multi-center, open-label, FIH study comprising of 2 study parts (Phase Ia, Phase Ib).

The Phase Ia (dose escalation) part of the study is designed to determine the safety, tolerability, and maximum tolerated dose (MTD)/recommended dose for expansion (RP2D) of BR101801 in subjects with relapsed/refractory B cell lymphoma, chronic lymphocytic leukemia (CLL)/small lymphocytic leukemia (SLL), and peripheral T cell lymphoma (PTCL).

The Phase Ib (dose expansion) part of the study is designed to assess tumor response and safety in specific advanced relapsed/refractory Peripheral T-cell lymphoma(PTCL) at a dose of BR101801 identified in Phase Ia. Once the RP2D has been determined in Phase Ia (dose escalation), Phase Ib (dose expansion) will commence.

DETAILED DESCRIPTION:
1. Phase Ia (Dose Escalation)

   Primary Objectives
   * To assess the safety and tolerability of BR101801 in patients with relapsed/refractory B-cell lymphoma, CLL/SLL, and PTCL.
   * To assess DLT and to determine the MTD and/or the RDE dose for BR101801 when administered orally on a daily schedule in 4-week cycles until disease progression.

   SecondaryObjectives
   * To characterize the plasma and urine PK of BR101801.
   * To assess the preliminary antitumor activity of BR101801.
2. Phase Ib (Dose Expansion)

Primary Objectives

• To assess the safety and tolerability of BR101801 at the RP2D dose in subjects with relapsed/refractory Peripheral T-cell lymphoma (PTCL).

SecondaryObjectives

* To assess clinical activity of BR101801 when administered orally on a daily schedule in 4-week cycles until disease progression.
* To assess the plasma PK of BR101801.

OUTLINE: This is a Phase I, multi-center, open-label, FIH study. The safety monitoring committee(SMC) will be responsible for safety oversight.

ELIGIBILITY:
<Inclusion Criteria>

1. Patients must sign an informed consent document
2. Female or male patients aged ≥ 18 years.
3. ECOG performance status ≤ 2.
4. Life expectancy more than 3 months.
5. Phase Ia:Patients with relapsed and/or refractory relapsed/refractory B-cell lymphoma, CLL/SLL, and PTCL diagnosed with World Health Organization (WHO) classification
6. Phase Ib: Subjects with PTCL NOS, PTCL AITL, Nodal PTCL with TFH and PTCL FTCL.
7. Patients have measurable disease based on the appropriate tumor type criteria( Phase Ib only)
8. Have a current need for systemic therapy, the assessment of the investigator.
9. An archival or fresh tumor tissue (ie, tissue block or series of at least 5 slides, up to 15 slides) is required and should be provided during the Screening Visit for Lymphoma subjects. Local review of pathology is required for study entry in Phase Ib only.
10. Phase Ia subjects should be prepared to undergo a fresh tumor biopsy during the study (tumor biopsies will be obtained from 1 to 2 subjects per cohort in Phase Ia).
11. Subject having laboratory values defined as:

    * Creatinine clearance (measured or calculated per institutional standard practice) ≥ 60 mL/min. GFR can also be used in place of creatinine clearance.
    * Total bilirubin < 1.5 × ULN, except for subjects with Gilbert's syndrome who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin < 1.5 × ULN.
    * ALT < 2.5 × ULN, except for subjects who have tumor involvement of the liver, who are included if ALT < 5 × ULN.
    * AST < 2.5 × ULN, except for subjects that have tumor involvement of the liver, who are included if AST < 5 × ULN.
    * Absolute neutrophil count > 1.0 × 109/L.
    * Platelet count > 75 × 109/L.
    * Hemoglobin > 8 g/dL.

<Exclusion Criteria>

1. Presence of overt leptomeningeal or active CNS metastases, or CNS metastases that require local CNS-directed therapy or increasing doses of corticosteroids within the prior 2 weeks. Patients with treated brain metastases should be neurologically stable and off steroids for at least 2 weeks before administration of any study treatment.
2. Impaired cardiac function or clinically significant cardiac disease
3. Patients with interstitial pneumonia or history of drug-induced interstitial pneumonia/pneumonitis.
4. Human immunodeficiency virus (HIV) infection.
5. Patients who are positive for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (HCVAb).
6. Chronic liver disease or chronic hepatitis
7. Any gastrointestinal disorders interfering with study drug absorption or are unable to swallow tablets or capsules.
8. Malignant disease, other than that being treated in this study.
9. Prior PI3K inhibitor will be accepted in the dose escalation part of the study (Phase Ia) only.
10. For patients with lymphoma:

    * Systemic antineoplastic therapy (including cytotoxic chemotherapy, alfa-interferon [INF], and toxin immunoconjugates) or any experimental therapy within 3 weeks or 5 half lives, whichever is shorter, before the first dose of study treatment.
    * Therapy with tyrosine kinase inhibitor within 5 half-lives before the first dose of study treatment.
    * Unconjugated monoclonal antibody therapies < 6 weeks before the first dose of study treatment.
11. Patients receiving systemic chronic steroid therapy or any immunosuppressive therapy (≥ 10 mg/day prednisone or equivalent).
12. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
13. Use of hematopoietic colony-stimulating growth factors, thrombopoietin mimetics, or erythroid-stimulating agents ≤ 2 weeks prior to start of study drug.
14. Patients with a history of stroke or having active neurological symptoms, with the exception of chronic conditions which, in the opinion of the neurologist, Investigator, and the Sponsor, would not impact ongoing neurologic assessments while on study treatment.
15. Active infection requiring systemic or antiviral antibiotic therapy.
16. Subjects with active CMV infection.
17. Subjects receiving moderate or potent CYP3A4 inhibitors or inducers and are unable to withdraw until 2 weeks or 5 times longer than the half-life, whichever is shorter, before the first dose of study treatment.
18. Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
19. Radiotherapy within 2 weeks of the first dose of study treatment, except for palliative radiotherapy to a limited-field, such as for the treatment of bone pain or a focally painful tumor mass.
20. Presence of CTCAE ≥ Grade 2 toxicity (except alopecia, peripheral neuropathy, and ototoxicity, which are excluded if ≥ CTCAE Grade 3) due to prior cancer therapy.
21. Participation in an interventional, investigational study within 2 weeks or 5 half-lives, whichever is shorter, of the first dose of study treatment.
22. Any medical condition that would, in the Investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns, compliance with clinical study procedures, or interpretation of study results.
23. Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
To determination of the MTD and RDE based on DLTs during Cycle 1 (Phase Ia) | From baseline to Week 4
  The recommended dose is determined by the number of patients who experience a dose limiting toxicity (DLT).
Number of participants with adverse events (AE) as a measure of safety and tolerability of BR101801 when administered at the MTD or recommended dose (Phase Ia and Ib) | through study completion, and about average of 1 year
  To evaluate safety and tolerability the aggregate review will include but is not limited to:
  * CTCAE TEAEs, treatment-related TEAEs, Grade 3 or higher TEAEs, Grade 3 or higher treatment-related TEAEs, serious treatment-related TEAEs, and TEAEs leading to death.
  * Laboratory results;
  * Vital signs;
  * ECGs;
  * Physical examination
  * ECOG performance status

SECONDARY OUTCOMES:
Cmax | Cycle1( each cycle is 28 days) Day 1 and Cycle 1( each cycle is 28 days) Day 15
  Maximum concentration obtained directly from the observed concentration versus time data.
AUC(0-inf) | Cycle1( each cycle is 28 days) Day 1
  Area under the plasma concentration-time curve from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation
AUC(0-last) | Cycle1( each cycle is 28 days) Day 1 and Cycle 1( each cycle is 28 days) Day 15, Pre-dose to 24 hours after dosing
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
AUC(0-tau) | Cycle1( each cycle is 28 days) Day 1 and Cycle 1( each cycle is 28 days) Day 15, dosing interval: 24 or 12 hours
  Area under the plasma concentration-time curve from time zero during a dosing interval
Ae | Cycle 1( each cycle is 28 days)Day 15, Pre-dose to 12 hours for BID dosing and Pre-dose to 24 hours for QD dosing
  Cumulative amount of unchanged drug excreted in urine

CONTACTS AND LOCATIONS:
Overall Officials: TM Kim, M.D, Ph.D, Principal Investigator — Seoul National University Hospital; SJ Kim, M.D, Ph.D, Principal Investigator — Samsung Medical Center; DH Yoon, M.D, Ph.D, Principal Investigator — Asan Medical Center; Jorge Chaves, M.D, Ph.D, Principal Investigator — Northwest Medical Specialities, PLLC; Emily Curran, M.D, Ph.D, Principal Investigator — University of Cincinnati; JS Kim, M.D, Ph.D, Principal Investigator — Severance Hospital, Yonsei University Health System; EY Lee, M.D, M.S, Principal Investigator — National Cancer Center; JO Lee, M.D, Ph.D, Principal Investigator — Seoul National University Bundang Hospital; DH Yang, M.D, Ph.D, Principal Investigator — Chonnam National University Hospital; WS Lee, M.D, Ph.D, Principal Investigator — Inje University
Locations (9):
- Henry Ford Hospital, Detroit, Michigan, United States
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Inje University Busan Paik Hospital, Busan
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul national university hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No